CLINICAL TRIAL: NCT07177287
Title: The Effect of a Navigator Nurse- Supported Mobile Application Developed Based on the IMB Model on the Quality of Life of Patients With Celiac Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, İlknur Bodur, Research Nurse / MSN (Master of Science in Nursing), Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IMB-CELIAC-QOL-2025-1
Record Dates: First submitted 2025-09-10; First posted 2025-09-16 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Celiac Disease; Adults With Celiac Disease
Keywords: quality of life; navigator nurse; mobile application; IMB model
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Navigator nurse-supported mobile application (IMB Model) (Experimental): Participants receiving the navigator nurse-supported mobile application based on the IMB model.
  Interventions: Behavioral: IMB navigator app
- Control: Standard care without mobile application (No Intervention): Participants receiving standard care without the mobile application.

INTERVENTIONS:
Behavioral: IMB navigator app — Mobile application developed based on the IMB model, supported by a navigator nurse. Includes educational content, reminders and behavioral support. Patients will be followed for 6 months.
  Arms: Experimental: Navigator nurse-supported mobile application (IMB Model)

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a navigator nurse-supported mobile application, developed based on the Information-Motivation-Behavioral Skills (IMB) model, on the quality of life of adult patients newly diagnosed with celiac disease. Participants will be randomized into intervention and control groups. The intervention group will use the mobile application with navigator nurse support for six months, while the control group will receive routine clinical education. Outcomes will be assessed through validated questionnaires and clinical data.

DETAILED DESCRIPTION:
Celiac disease is an autoimmune disorder characterized by gluten intolerance, leading to intestinal mucosal damage and a variety of physical and psychological symptoms. Strict adherence to a gluten-free diet remains the only effective treatment but is challenging due to hidden gluten sources and limited knowledge.

The IMB model provides a theoretical framework suggesting that health-related behaviors are influenced by information, motivation, and behavioral skills. A navigator nurse can support patients by providing education, motivation, and personalized guidance.

In this study, a mobile application was developed to provide education and continuous support to celiac patients under the guidance of a navigator nurse. The study hypothesizes that this intervention will improve health-related quality of life compared to standard clinical education.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Newly diagnosed with celiac disease
* Owning a smartphone and able to use the application
* Able to speak and understand Turkish
* Voluntary participation (informed consent)

Exclusion Criteria:

* Severe gluten hypersensitivity
* Failure to meet inclusion criteria
* Withdrawal of consent during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Improving the quality of life of celiac patients | 6 months
  Change in quality of life scores measured by a validated questionnaire for celiac disease patients (e.g., Celiac Disease Quality of Life Survey) from baseline to the end of the intervention.
  Health-Related Quality of Life Questionnaire in Celiac Disease: The questionnaire was developed by Hauser et al. and validated in Turkey by Aksan et al. It assesses how adult celiac patients have felt over the past two weeks by asking about disease-related symptoms, general well-being, and emotional state. The questionnaire consists of 28 items, evaluated across four subscales: emotional, social, gastrointestinal, and worries. Each item is rated on a 7-point Likert scale. Participants can score a minimum of 0 and a maximum of 49 points in each subscale. The total score ranges between 0 and 196, with lower scores reflecting lower quality of life.

SECONDARY OUTCOMES:
Adherence to Gluten-Free Diet | 6 months
  Measurement Tool: Self-reported adherence and dietary records. Outcome Metric: Percentage of adherence (%0-100).
Patient Motivation Level | 6 months
  Measurement Tool: Motivation Assessment Tool (developed by the investigator based on literature review; validated by Content Validity Index [CVI]).
  Outcome Metric: Item-based evaluation; mean score will be calculated for each item, and higher mean values will indicate greater motivation.
Patient Engagement with the Mobile Application | 6 months
  Measurement Tool: In-app communication records (number of questions asked to the navigator nurse, number of forum posts/replies).
  Outcome Metric: Average number of patient-initiated questions and forum interactions per month.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal TÜZER, Study Director — Faculty of Health Sciences, Ankara Yıldırım Beyazıt University
Locations (1):
- Ankara Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No